CLINICAL TRIAL: NCT04763785
Title: Development of a Keratoconus Detection Algorithm by Deep Learning Analysis and Its Validation on Eyestar Images
Acronym: DKDA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: DKDA-E900-2020
Record Dates: First submitted 2021-02-14; First posted 2021-02-21 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-06

CONDITIONS: Keratoconus; Eye Diseases; Cataract; Corneal Ectasia
Keywords: Keratoconus; Eye Diseases; Cataract; Corneal Imaging; Corneal Topography; Corneal Tomography; Corneal Ectasia
MeSH Terms: conditions — Keratoconus; Eye Diseases; Cataract | interventions — Biometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with keratoconus corneas: Corneal tomography on patients with keratoconus diagnosis
  Interventions: Device: Corneal tomography with Eyestar 900; Device: Corneal tomography with Pentacam; Device: Biometry with IOL-Master
- participants with healthy corneas: Corneal tomography on healthy participants
  Interventions: Device: Corneal tomography with Eyestar 900; Device: Corneal tomography with Pentacam; Device: Biometry with IOL-Master
- retrospective part: fully anonymised Picture data of existing 4500 patients
  Interventions: Other: retrospective analysis, no intervention

INTERVENTIONS:
Device: Corneal tomography with Eyestar 900 — Non-invasive corneal tomography to develop an imaging analysis algorithm for keratoconus corneas
  Groups: Patients with keratoconus corneas; participants with healthy corneas
Device: Corneal tomography with Pentacam — Non-invasive corneal tomography to develop an imaging analysis algorithm for keratoconus corneas
  Groups: Patients with keratoconus corneas; participants with healthy corneas
Device: Biometry with IOL-Master — Non-invasive biometry for presurgical intraocular lens calculation
  Groups: Patients with keratoconus corneas; participants with healthy corneas
Other: retrospective analysis, no intervention — retrospective analysis of 4500 existing, fully anonymised picture data
  Groups: retrospective part

SUMMARY:
Monocentric clinical study to develop an imaging analysis algorithm for the Eyestar 900 to identify keratoconus corneas and improve biometry for intraocular lens calculations

DETAILED DESCRIPTION:
Keratoconus is a progressive corneal ectatic disorder, characterised by thinning, protrusion and irregularity. Corneal imaging is crucial in keratoconus detection and progression analysis. Detection of keratoconus in early stages is important and has therapeutic consequence, whether to plan a surgical intervention or calculating an intraocular lens, before cataract surgery, as standard lens calculation techniques may lead to wrong results in patients with a keratoconus.

The Eyestar 900 is a swept-source OCT biometer and has the potential to be used for early keratoconus identification and progression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with all stages of keratoconus
2. Patients with healthy corneas

Exclusion Criteria:

1. Keratoconus patients with hydrops, status following hydrops
2. Patients with degenerative corneal diseases
3. Patients after corneal surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: retrospective part: anonymised picture-data of 4500 patients prospective part: 150 keratoconus patients and 150 healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 4800 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Keratoconus identification | 2.5 years
  Classification accuracy of the keratoconus identification algorithm for the Eyestar device in comparison to the gold standard (Belin-Ambrosio Enhanced Extasia Deviation Index) BAD_D in Pentacam images.

SECONDARY OUTCOMES:
Feasibility in clinical practice | 2.5 years
  Evaluation of the feasibility (percentage of valid measurements without errors and/or problems in image aquisition) of cornea measurements in keratoconus and healthy eyes.

CONTACTS AND LOCATIONS:
Overall Officials: Früh Beatrice, Prof.Dr. med., Principal Investigator — Universitätsklinik für Augenheilkunde, Inselspital Bern
Locations (1):
- Universitätsklinik für Augenheilkunde, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No